CLINICAL TRIAL: NCT01721226
Title: CARE Corrections: Technology for Jail HIV/HCV Testing, Linkage, and Care (TLC)
Acronym: CARE+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: The Miriam Hospital (Other); New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01DA030747-01 (NIH)
Record Dates: First submitted 2012-10-16; First posted 2012-11-05 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Human Immunodeficiency Virus
Keywords: Linkage to HIV care following release from prison; Anti-retroviral therapy adherence after release from prison; HIV loads after release from prison; information technology and ART adherence; information technology and linkage to HIV care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Sham Comparator): Participants in the Control Arm will receive standard discharge services according to the standards of care for that facility. In addition, participants in this arm will view an educational video on opiate overdose prevention. Study participants in the Control Arm will be followed after release/study enrollment, just like participants in the Intervention Arm, and Plasma Viral Loads will be collected from them at baseline and follow-up.
  Interventions: Other: Educational video on opiate overdose prevention
- CARE tool and cell phone/text messaging (Experimental): The Intervention Arm will complete the CARE tool device, a technology based HIV-counseling tool, and will receive text message reminders about HIV medical appointments and the importance of taking HIV medications. Study participants in this arm will be followed after release/study enrollment, just like participants in the Control Arm, and Plasma Viral Loads will be collected from them at baseline and follow-up.
  Interventions: Device: Intervention Arm (computer-based CARE+ Corrections tool)

INTERVENTIONS:
Device: Intervention Arm (computer-based CARE+ Corrections tool) — Study participants in the intervention arm will complete the computer-based CARE+ Corrections tool at baseline. The CARE tool provides tailored feedback based on the participants' responses to a series of questions included in the counseling session. Participants in this arm of the study recruited inside the DC DOC will receive typical discharge planning services as conducted by the correctional facility. Participants will be followed for six months after release/study enrollment. At the post-release baseline visit, participants in the intervention arm will receive a cell phone/SMS text messaging intervention consisting of using cell phone-delivered SMS text messages with the intent of improving linkage to community HIV care and adherence to ART (if prescribed.)
  Arms: CARE tool and cell phone/text messaging
Other: Educational video on opiate overdose prevention — Participants in the Control Arm will view an educational video on opiate overdose prevention in jail prior to release. Control arm participants will be followed after release/study enrollment, just like participants in the Intervention Arm, and Plasma Viral Loads will be collected from them at baseline and follow-up.
  Arms: Control Arm

SUMMARY:
The purpose of this study is to determine whether an intervention (CARE+ Corrections) delivered to HIV-infected detainees within the DC Department of Corrections (DOC) and recently -released ex-detainees in the community can improve linkage to community HIV care and adherence to HIV medications after release, and ultimately achieve or maintain HIV viral suppression following community re-entry.

DETAILED DESCRIPTION:
The intervention is modeled after CARE, a technology based HIV-counseling tool used in other settings. The investigators have adapted CARE to create CARE+ Corrections, a tool designed specifically for incarcerated and recently-released populations. New and innovative information communication tools (ICT), including a cell phone/text messaging component delivered in the community after release from jail, will be included in the intervention.

The study is a randomized controlled trial. One half of the participants will receive the intervention either inside the jail, in addition to standard discharge planning services, or in the community right after release. The other half of the participants will view an educational video related to the prevention of drug overdose following release, in addition to standard discharge planning services, or in the community right after release. The investigators will follow all participants for 6 months post release/study enrollment and determine if the linkage to community care and adherence to HIV medications was higher in the intervention arm.

The study also has an evaluation component to it. The evaluation component consists in a series of qualitative interviews with the goal of gaining a better understanding of the barriers and facilitators involved in implementing the CARE+ Corrections intervention and to better assess the usability and participants' experiences with the CARE+ Corrections intervention. The semi-structured interviews are being conducted among the following groups: 1) managers and staff at local correctional facilities and agencies which have interaction with HIV+ individuals transitioning to the community; 2) leadership and selected staff at relevant and targeted community-based organizations; and 3) selected study participants from the intervention group of the RCT. the interviews elicit perspectives on the foreseen facilitators and challenges in implementing the CARE+ Corrections tool at their respective organizations as well as their perception on the acceptability of the tool. We also ask their views about the intervention and the post-release experiences of HIV-positive individuals who complete the CARE+ Corrections Tool and receive the text message plan.

No prisoners will be involved in this subsection of the study.

ELIGIBILITY:
Inclusion Criteria:

* Currently detained in jail or released from the jail/prison 6 months ago or less
* 18 years of age or older
* English speaking
* Able to provide informed consent for research participation
* Anticipated release from the DOC to the community (or living in the community if recently released ex-detainee)
* Confirmed to be HIV-infected by self-report
* Live in metropolitan Washington, DC area
* Able to read at 8th grade level as assessed by brief literacy screen

Exclusion Criteria:

* Expected release to restricted setting (or currently living in a restricted setting if recruited in the community), including residential drug treatment, sober house, half-way house, or similar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-08; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Kuo, PhD, MPH, Principal Investigator — George Washington University School of Public Health and Health Services
Locations (1):
- Family and Medical Counseling Services, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Uhrig Castonguay BJ, Cressman AE, Kuo I, Patrick R, Trezza C, Cates A, Olsen H, Peterson J, Kurth A, Bazerman LB, Beckwith CG. The Implementation of a Text Messaging Intervention to Improve HIV Continuum of Care Outcomes Among Persons Recently Released From Correctional Facilities: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Feb 13;8(2):e16220. doi: 10.2196/16220. PMID 32053119
- [Derived] Beckwith C, Castonguay BU, Trezza C, Bazerman L, Patrick R, Cates A, Olsen H, Kurth A, Liu T, Peterson J, Kuo I. Gender Differences in HIV Care among Criminal Justice-Involved Persons: Baseline Data from the CARE+ Corrections Study. PLoS One. 2017 Jan 12;12(1):e0169078. doi: 10.1371/journal.pone.0169078. eCollection 2017. PMID 28081178

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Arm | CARE Tool and Cell Phone/Text Messaging
Started | 55 | 57
Baseline | 53 | 57
Week 12 | 48 | 53
Week 24 | 50 | 50
Completed | 50 | 50
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | CARE Tool and Cell Phone/Text Messaging | Total
Number analyzed (Participants) | 55 | 57 | 112
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 39 [30 to 57] | 42 [30 to 50] | 41.5 [30 to 49]
Sex/Gender, Customized [Number; unit: participants]
  Male | 32 | 33 | 65
  Female | 13 | 14 | 27
  Transgender | 10 | 10 | 20
Baseline Viral Suppression [Number; unit: participants]
  Virally suppressed (PVL<100) | 37 | 32 | 69
  Not virally suppressed (PVL >=100) | 17 | 22 | 39

OUTCOME MEASURES:

1. Primary Outcome: Plasma Viral Load Suppression
Description: Plasma viral load at 24 weeks measured by viral load testing or medical chart abstraction
Time Frame: 24 weeks
Population: All study participants with available PVL data
Measure: Number; unit: participants
Arm/Group | Control Arm | CARE Tool and Cell Phone/Text Messaging
Number analyzed (Participants) | 49 | 47
participants
  Virally suppressed (PVL<100) | 26 | 23
  Not virally suppressed (PVL >=100) | 23 | 24

2. Secondary Outcome: Linkage to Community Care
Description: At least 1 visit to health care provider in past 24 weeks/6 months
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | CARE Tool and Cell Phone/Text Messaging
Number analyzed (Participants) | 51 | 52
Participants
  Yes-achieved outcome | 45 | 47
  No-did not achieve outcome | 6 | 5

ADVERSE EVENTS:
Time Frame: Enrollment and follow-up period
Arm/Group | Control Arm | CARE Tool and Cell Phone/Text Messaging
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/57
Other Adverse Events (participants affected / at risk) | 0/55 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No